CLINICAL TRIAL: NCT05033171
Title: The Changing of the Fixation-rod Shape After Posterior Correction Segmentdesis in Adolescent Idiopathic Scoliosis
Brief Title: Rod Shape Changing After Scoliosis Correction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP-CC-Ortho-RodShape
Record Dates: First submitted 2021-08-29; First posted 2021-09-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Scoliosis Idiopathic; Scoliosis, Severe
Keywords: scoliosis; posterior segmentdesis; 3D scanning; EOS 2D/3D
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with scoliosis induced surgical indication (Cobb-degree>45).
  * Posterior screw-rod fixation segmentdesis
  * Before the implantation, right after the implantation and after the in situ bending 3D scanning of the rod using Artec Eva Spider type manual 3D scanner will be performed. Scanning is possible from a more than 60 cm distance, so that means the operational area stays sterile.
  * EOS Micro Dose imaging will be done on the third day after surgery, on the third, the sixth, the twelfth and twenty fourth month after surgery (as in the actual clinical protocal).
  Interventions: Diagnostic Test: 3D Scanning; Diagnostic Test: EOS 2D/3D scanning

INTERVENTIONS:
Diagnostic Test: 3D Scanning — 3D scanning of the rod using Artec Eva Spider type manual 3D scanner
Diagnostic Test: EOS 2D/3D scanning — EOS Micro Dose imaging will be done on the third day after surgery, on the third, the sixth, the twelfth and twenty fourth month after surgery.

SUMMARY:
The change of the fixation-rod after posterior srew-rod fixation segmentdesis is not widely known. The recent development of the 3D scanning technics and the opportunities of the EOS 2D/3D system made us possible to have the exact rod shape immediately after implantation, and at each control examination. These progressions made us available to follow up the shape changing of the fixation-rod, hereby the changing of the correction.

DETAILED DESCRIPTION:
The adolescent idiopathic scoliosis can affect the 0,5-2% of the European population. One of the widely accepted treatment of severe scoliosis (Cobb angle is over 40-50°, or more than 10° progression observed a year) is posterior correction segmentdesis with screw and rod instrumentation. As a scoliosis treatment center, about 90-110 scoliosis correction surgeries are performed in our department, using conventional preoperative planning, coronal and sagittal translation technique from posterolateral approach.

An EOS 2D/3D system is available in our department making possible the scanning of the patient with upright biplanar ultra-low dose x-rays technique. The SterEOS software makes us possible to reconstruct the surface of the spine, pelvis and lower limb. The biplanar modality of the images makes possible to 3D reconstruct any simple shape using CAD (computer-aided design) softwares.

The recent updates in the 3D scanning technology also made us possible to perform intraoperative scannings without harming the sterility.

The aim of the study to define the change of the fixation-rod's shape after scoliosis correction surgery.

Main hypothesis: there is significant change in the rod shape after implantation

Secondary hypothesis 1: during the implant of the rod, it will loose from the prebent correction depending of the severity and rigidity of the curve.

Secondary hypothesis 2: in the early stage of the rehabilitation, after the mobilization the shape of the rod (and the spinal parameters) can change Secondary hypothesis 3: after the 3. month postoperatively the shape of rod does not change anymore

ELIGIBILITY:
Inclusion Criteria:

* routine patient care of University of Pécs Medical School Department of Orthopaedics
* diagnosed idiopathic adolescent scoliosis
* scoliosis induced surgical indication (Cobb-degree>45)

Exclusion Criteria:

* early onset or adult degenerative scoliosis
* scoliosis with known origin
* the angle of the curve does not reach the criteria of surgical indication (Cobb-degree<45)
* former spine surgery

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Shape changing of the rod | 2 years
  The fitted 3D models of the implanted rod right after implantation, 3 day, than 3-6-12-24 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Than, PhD, Study Chair — UP MS Department of Orthopaedics
Locations (1):
- Ádám Schlégl, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No